CLINICAL TRIAL: NCT03436303
Title: The Effect and Risk of Conjugated Estrogens Combined With Different Types of Progestin in the Treatment of Menopause Syndrome During Window Phase
Brief Title: The Benefits and Risks of Different Menopausal Hormone Replacement Therapy Regimes in the Treatment of Menopause Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Aijun Sun, professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRT14021808
Record Dates: First submitted 2018-02-02; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Menopause Syndrome
Keywords: Menopause Syndrome; low dose estrogen; progestin
MeSH Terms: interventions — 2-chloroethyl ethyl sulfide; Dydrogesterone

STUDY DESIGN:
Intervention Model Description: randomly assigned to three groups: CEE 0.3 mg/micronized progesterone (MP) 100 mg group, CEE 0.625 mg/MP 100 mg group,CEE 0.625 mg/dydrogesterone 10 mg group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CEE 0.625 mg/MP 100mg (Experimental): CEE 0.625 mg/micronized progesterone (MP) 100 mg daily for the last 12 days of every 28 days for two years
  Interventions: Drug: CEE 0.625 mg/MP 100mg
- CEE 0.3 mg/MP 100mg (Experimental): CEE 0.3mg/micronized progesterone (MP) 100 mg daily for the last 12 days of every 28 days for two years
  Interventions: Drug: CEE 0.3 mg/MP 100mg
- CEE 0.625 mg/dydrogesterone 10mg (Experimental): CEE 0.625 mg/dydrogesterone 10 mg daily for the last 12 days of every 28 days for two years
  Interventions: Drug: CEE 0.625mg/dydrogesterone

INTERVENTIONS:
Drug: CEE 0.625 mg/MP 100mg — CEE 0.625 mg daily/MP 100mg daily for the last 12 days of every 28 days for two years
  Arms: CEE 0.625 mg/MP 100mg
Drug: CEE 0.3 mg/MP 100mg — CEE 0.3 mg daily/MP 100mg daily for the last 12 days of every 28 days for two years
  Arms: CEE 0.3 mg/MP 100mg
Drug: CEE 0.625mg/dydrogesterone — CEE 0.3 mg/dydrogesterone 10mg daily for the last 12 days of every 28 days for two years
  Arms: CEE 0.625 mg/dydrogesterone 10mg

SUMMARY:
A prospective, open-label, randomized controlled clinical trial to compare the benefits and risks of half-dose or standard-dose conjugated equine estrogens(CEE) plus natural progesterone or dydrogesterone in menopausal hormone therapy .

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized controlled clinical trial compare the benefits and risks of half-dose or standard-dose conjugated equine estrogens(CEE) plus natural progesterone or dydrogesterone in menopausal hormone therapy during window phase. 120 Healthy postmenopausal women with intact uterus seeking treatment for menopausal symptoms are enrolled in this study.Participants are randomized into three groups, the CEE 0.3 mg/micronized progesterone (MP) 100 mg group; CEE 0.625 mg/MP 100 mg group; CEE 0.625 mg/dydrogesterone 10 mg group,metabolic parameters,body composition,bone mineral density,breast cancer risk factors and life quality will be measure at baseline,one year and two year intervention.The investigators hypothesize there may be differences of these parameters measured among three groups after intervention.

ELIGIBILITY:
Inclusion Criteria:

1. 40 and 60 years old;
2. natural amenorrhea for more than 6 months but less than 5 years;
3. suffered by menopause symptoms and seeking for treatment;
4. serum follicle-stimulating hormone levels >40 IU/L and serum estradiol <30 pg/ml.

Exclusion Criteria:

1. contraindications for menopausal hormone therapy;
2. complications including: uterine myoma more than 3 centimeter in diameter, endometriosis, uncontrolled hypertension or diabetes mellitus, thromboembolic disease history or high risk for developing thromboembolic disease, epilepsy, asthma, hyperprolactinemia, first degree relative has breast cancer;
3. cardiovascular, chronic liver, thyroid or kidney diseases; a history of cancer; a disease or condition that could influence the participants' ability to follow the study protocol;
4. alcohol or drug abuse within the last 3 months;
5. use of hormone therapy in the past 3months;
6. endometrial thickness more than 5mm even after progestin withdrawal;
7. abnormal cervical scraping smear;
8. allergic to any ingredient of the drugs;
9. participation in other clinical trials within the last 6 months.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 120 (Estimated)
Dates: Start 2014-02-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
LDL-cholesterol | 5 minutes
body fat mass percentage | 5 minutes
  DEXA method
breast mammography | 5 minutes

SECONDARY OUTCOMES:
glucose | 5 minutes
bone mineral density | 5 minutes
Mini-mental State Examination score | 5 minutes
  Questionnaire.The score range is 0-30.Total score greater than or equal to 24 points indicates a normal cognition,below this, scores can indicate cognitive impairment.
HAD scale | 5 minutes
  questionnaire to evaluate anxiety and depression.The total score is 0-20.Total score 0-7 is normal,8-10 maybe borderline anxiety or depression,11-20 indicates obvious anxiety or depression.
modified Kupperman score | 5 minutes
  questionnaire to evaluate the menopause symptom.The total score range is 0-63.Total score below 6 is normal,6-15 is mild,16-30 is moderate, above 30 is severe
Endometrial thickness | 5 minutes
  ultrasound
weight | 5 minutes
serum creatinine | 5 minutes
serum glutamic pyretic transaminase | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Aijun Sun, MD, Principal Investigator — Peking Union Medical College Hospital,Peking Union Medical College, Chinese Academy of Medicine Sciences
Locations (1):
- Lei Li, Beijing, China/Beiing, China

IPD SHARING:
Plan to Share IPD: Yes
Network platform, and the website will be attached later.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Within 2 months after the trial complete
Access Criteria: Data access requests will be reviewed by an external independent review panel.Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Thorneycroft IH, Lindsay R, Pickar JH. Body composition during treatment with conjugated estrogens with and without medroxyprogesterone acetate: analysis of the women's Health, Osteoporosis, Progestin, Estrogen (HOPE) trial. Am J Obstet Gynecol. 2007 Aug;197(2):137.e1-7. doi: 10.1016/j.ajog.2007.05.042. PMID 17689624
- [Background] Margolis KL, Bonds DE, Rodabough RJ, Tinker L, Phillips LS, Allen C, Bassford T, Burke G, Torrens J, Howard BV; Women's Health Initiative Investigators. Effect of oestrogen plus progestin on the incidence of diabetes in postmenopausal women: results from the Women's Health Initiative Hormone Trial. Diabetologia. 2004 Jul;47(7):1175-1187. doi: 10.1007/s00125-004-1448-x. Epub 2004 Jul 14. PMID 15252707